CLINICAL TRIAL: NCT06750783
Title: A Randomized Controlled Study on the Effects of Xuezhikang and Atorvastatin on Blood Glucose and Lipid Levels in Patients With Dyslipidemia and Prediabetes
Brief Title: The Effects of Xuezhikang and Atorvastatin on Lipid in Patients With Dyslipidemia and Prediabetes
Acronym: Xuezhikang
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.0 20240725
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-12

CONDITIONS: Prediabetic State (IGT)
Keywords: XUEZHIKANG; atorvastatin; glucose metabolism; blood glucose fluctuations; diabetes
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus | interventions — xuezhikang; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin group (Experimental): According to routine clinical practice, patients with dyslipidemia with prediabetes were given atorvastatin at a dose of 20 mg qd；
  Interventions: Drug: Atorvastatin
- Xuezhikang group (Experimental): The Xuezhikang group takes Xuezhikang at a dose of 600 milligrams twice a day, orally after meals;
  Interventions: Drug: Xuezhikang

INTERVENTIONS:
Drug: Xuezhikang — The Xuezhikang group takes Xuezhikang at a dose of 600 milligrams twice a day, orally after meals;
  Arms: Xuezhikang group
Drug: Atorvastatin — The atorvastatin group takes atorvastatin 20mg once a day, orally after meals.
  Arms: Atorvastatin group

SUMMARY:
This study compares the impact of Xuezhikang and atorvastatin on glucose metabolism to explore the incidence of prediabetes patients developing diabetes after 24 weeks of Xuezhikang use, and by investigating the effect of Xuezhikang on blood glucose fluctuations, discusses the possible mechanisms by which Xuezhikang affects glucose metabolism.

DETAILED DESCRIPTION:
The development of chronic complications of diabetes is not only closely related to HbA1c, but may also correlate with blood glucose fluctuations, and the mechanisms may be related to including oxidative stress, inflammation, endothelial dysfunction, and altered gene expression. Glycemic fluctuations are not only important in diabetic patients, but also in prediabetic patients where changes have already been observed. Intraday glucose fluctuations in patients with abnormal glucose tolerance are already significantly higher, up to 50% higher than in those with normal glucose regulation. The study of blood glucose fluctuation and pancreatic function found that the level of blood glucose fluctuation in normal glucose regulators, pre-diabetic and gestational diabetic patients was negatively correlated with early phase insulin secretion function, indicating that those with large blood glucose fluctuation have relatively poor pancreatic function, suggesting that early changes in pancreatic function can affect blood glucose fluctuation. Therefore, the authors believe that blood glucose fluctuation may be significant for the progression of pre-diabetes to diabetes, and can be used for early warning of diabetes. In this study, we investigated the lipid-lowering effect of the natural lipid-regulating drug Lipotecan and its effect on insulin resistance, blood glucose fluctuation and new-onset diabetes in patients with dyslipidemia with prediabetes.

This is a multicenter, prospective, open-label, superiority randomized controlled study to explore the effects of applying Lipitor (dose 600mg bid) versus atorvastatin (20mg qd) on the incidence of new-onset diabetes mellitus, glucose fluctuation, and the differences in the pre and post changes in lipid profiles in patients with dyslipidemia with pre-diabetes mellitus, respectively.

All subjects were informed and the study was intended to be approved by the Ethics Committee of Beijing Tsinghua Changgeng Hospital, Tsinghua University.

Hypothesis: Patients with prediabetes combined with dyslipidemia were orally administered Lipitor (600 mg bid).The rate of new-onset diabetes is lower than that of atorvastatin (200 mg qd) treatment group.

The Lipocon group will receive Lipocon at a dose of 600mg twice daily with meals, and the Atorvastatin group will receive Atorvastatin 20mg once daily orally with meals.All patients will be treated for 24 weeks. Patients are not allowed to use other lipid-lowering medications throughout the study period.

All subjects will be required to take a cell phone related medical history, including general condition, past medical history, current medical history and history of drug use. The laboratory collected blood specimens from the subjects in accordance with the clinical diagnosis and treatment, tested glycated hemoglobin, glucose, insulin and c-peptide by oral glucose tolerance test in fasting, 0.5h, 1h and 2h after sugar water, and monitored the basic liver function, renal function, lipid profile and creatine kinase of all subjects, and the venous blood taken was strictly verified by the laboratory departments of the respective centers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* No gender restrictions;
* Definition of pre diabetes: All subjects were tested with 75g OGTT to measure fasting and 2h venous serum glucose and glycosylated hemoglobin. Fasting blood glucose ≥ 6.1 and < 7mmol/L, 2-hour serum glucose ≥ 7.8 and < 11.1mmol/L after glucose load, and glycated hemoglobin<6.5%;
* Abnormal lipid metabolism: LDL-c ≥ 3.4 mmol/L and<4.9 mmol/L, and TG ≤ 5.6 mmol/L; (2) Non-HDL-c ≥ 4.1mmol/L and<5.7 mmol/L, and TG ≤ 5.6 mmol/L;
* Voluntarily sign the informed consent form.

Exclusion Criteria:

* Patients who have met the diagnosis of diabetes;
* Within 3 months prior to signing the informed consent form, there was an acute coronary syndrome, stroke, or transient ischemic attack.
* ALT/AST>3 times ULN;
* Known myopathy, rhabdomyolysis, or creatine kinase levels greater than 4-fold ULN, and not caused by muscle injury;
* Pregnant or planning to conceive;
* Have used any lipid-lowering drugs within 3 months;
* Individuals with allergies/contraindications to Xuezhikang and Atorvastatin.
* Suffering from any of the following diseases: uncontrolled hyperthyroidism and hypothyroidism, severe heart failure, malignant tumors, hematopoietic system diseases, digestive system diseases affecting digestion and/or absorption function, mental disorders, other serious or unstable physical diseases.
* History of alcohol or drug abuse or dependence within 3 months prior to joining the trial.
* Participated in clinical trials of other drugs or devices within 3 months prior to joining the trial.
* Researchers believe that other situations are not suitable for participating in the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of diabetes | 24 weeks
  Collect blood samples from subjects, measure patients' glycated hemoglobin, and detect blood glucose levels at fasting, 0.5 hours, 1 hour, and 2 hours after drinking 75g glucose water through the oral glucose tolerance test (OGTT) (the time is calculated from the start of drinking the glucose water).

CONTACTS AND LOCATIONS:
Overall Officials: lixia jin, phD, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (3):
- China (3):
  - Beiqijia Community Health Service Center, Changping District, Beijing, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Xiaotangshan Community Health Service Center, Changping District, Beijing, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No